CLINICAL TRIAL: NCT02490787
Title: A Multi-centre, Randomised, Placebo Controlled, Double Blinded, Multiple Dose Trial Investigating Safety, Pharmacokinetics and Pharmacodynamics of Concizumab Administered Subcutaneously to Haemophilia A Subjects (Explorer™3)
Brief Title: Trial Investigating Safety, Pharmacokinetics and Pharmacodynamics of Concizumab Administered Subcutaneously to Haemophilia A Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN7415-4159; 2014-003793-16 (EudraCT Number); U1111-1161-1501 (Other: WHO); NL53826.018.15 (Registry Identifier: Netherlands Registry)
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — concizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concizumab (Experimental)
  Interventions: Drug: Concizumab; Drug: placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Concizumab — Administered subcutaneously (s.c., under the skin) at five different dose levels (ranging from 0.25 to 1.5 mg/kg)
  Arms: Concizumab
Drug: placebo — Administered subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate safety, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of concizumab administered subcutaneously to haemophilia A subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects diagnosed with haemophilia A without inhibitors present at screening and currently treated on-demand
* Subjects with a baseline level of factor VIII below or equal to 2 % based on medical records
* Age between 18 and 64 years both inclusive, at the time of signing informed consent
* Body weight between 50 and 100 kg, both inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products
* Platelet count below 50x10^9/L at screening
* Any clinical signs or known history of thromboembolic events, or subjects considered at high risk of thromboembolic events as judged by the investigator
* Subjects at increased risk of cardiovascular disease as judged by the investigator

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | From first trial drug administration (day 1) to 11 weeks after the first trial product administration

SECONDARY OUTCOMES:
Trough level of concizumab | Prior to the last s.c. dose administration (day 42)
Frequency of binding non-neutralizing anti-concizumab antibodies | From first trial drug administration (day 1) to 11 weeks after the first trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (33):
- United States (8):
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Melbourne, Victoria
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Zagreb, Croatia
- France (3):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Rennes
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Homburg
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Malaysia (2):
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Kuching
- Netherlands (3):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Nijmegen
  - Novo Nordisk Investigational Site, Utrecht
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Novo Nordisk Investigational Site, Bornova-IZMIR, Turkey (Türkiye)
- Ukraine (2):
  - Novo Nordisk Investigational Site, Dnipropetrovsk
  - Novo Nordisk Investigational Site, Lviv
- United Kingdom (3):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Southampton

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com